CLINICAL TRIAL: NCT00674167
Title: The Effect of Preoperative Docetaxel, Cisplatin and Capecitabine on Serum RUNX3 Hypermethylation Status in Patients With Gastric and Lower Oesophagus Adenocarcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Dr. Yong Wei Peng, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA02/33/06; 2006/00462 (Other: NHG Domain Specific Review Boards); CTC0700084 (Other: Health Sciences Authority)
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Docetaxel (Experimental): Three cycles of chemotherapy will be administered before surgery with docetaxel and cisplatin at 30 mg/m² on day 1 and 8 in a 21 day treatment cycles.
  Interventions: Drug: Docetaxel
- Cisplatin (Experimental): Three cycles of chemotherapy will be administered before surgery with cisplatin at 30 mg/m² on day 1 and 8 in a 21 day treatment cycle.
  Interventions: Drug: Cisplatin
- Capecitabine (Experimental): Three cycles of chemotherapy will be administered before surgery with capecitabine at 750 mg/m² twice daily from day 1 to 14 in a 21 day treatment cycles.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxel — Three cycles of chemotherapy will be administered before surgery with docetaxel at 30 mg/m² on day 1 and 8 in a 21 day treatment cycles.
  Arms: Docetaxel
Drug: Cisplatin — Three cycles of chemotherapy will be administered before surgery with cisplatin at 30 mg/m² on day 1 and 8 in a 21 day treatment cycle.
  Arms: Cisplatin
Drug: Capecitabine — Three cycles of chemotherapy will be administered before surgery with capecitabine at 750 mg/m² twice daily from day 1 to 14 in a 21 day treatment cycle.
  Arms: Capecitabine

SUMMARY:
* To assess the radiological response, curative resection rate of preoperative docetaxel/cisplatin/capecitabine(DCX).
* To correlate treatment response with serum RUNX3 promoter hypermethylation.
* To determine the toxicities of preoperative DCX
* To determine the time to progression/overall survival of preoperative DCX

DETAILED DESCRIPTION:
Background:

Pre-operative chemotherapy down size and down stage tumours prior to surgery and improves treatment outcome. However, current chemotherapy regime requires long terrn venous access for protracted chemotherapy infusion. Despite encouraging response rate, there are still a substantial number who did not achieve curative resection after pre-operative chemotherapy. Hence there is a need to develop 1) a more convenient and effective regimen and 2) a surrogate for treatment response so that the non-responder can be identified early.

Specific aims:

To assess the radiological response, curative resection rate of preoperative docetaxel/cisplatin and capecitabine in patients with Stage II & III gastric or lower oesophageal adenocarcinoma and to correlate treatment response with serum RUNX3 methylation status.

Hypotheses:

We hypothesize that the proposed preoperative regimen is effective in gastric cancer and can be safely delivered. In addition, RUNX3 promoter hypermethylation status can be a surrogate for treatment response.

Methodology:

This is a phase II study design to assess the response and tolerability of preoperative docetaxel, cisplatin and capecitabine in patients with operable gastric cancer. Simon's two-stage design is used to calculate the sample size for this Phase II trial, using two levels of response rate, P0 (20%) and P1 (50%). Accordingly, 20 patients is required for this study; 8 patients will be accrued for the first stage followed by 12 more patients when three or more responses are observed during the first stage. The alpha level of the design is 0.04 and power is 0.86. Serum measurement of tumour's RUNX3 promoter hypermethylation will be performed prior to each treatment cycle to evaluate its role as a biomarker for treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the stomach or lower third of the oesophagusthat considered to be stage II (through the submucosa) or higher, with no evidence of distant metastases, or locally advanced inoperable disease, as evaluated by computed tomography, chest radiography, ultrasonography, or laparoscopy.
* Patients must have evaluable or measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan.
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of DCX in patients <18 years of age, children are excluded from this study.
* ECOG performance status <= 1 (see Appendix A).
* Patients must have normal organ and marrow function as defined below:

X leukocytes >= 3,000/mcL X absolute neutrophil count >= 1,500/mcL X platelets >= 100,000/mcL X total bilirubin within normal institutional limits X AST(SGOT)/ALT(SGPT) <= 2.5 X institutional upper limit of normal X creatinine within normal institutional limits

* The effects of DCX on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had prior chemotherapy or radiotherapy.
* Patients may not be receiving any other investigational agents.
* Patients with stage I or IV cancer of the stomach or lower oesophagus.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetacel, cisplatin or capecitabine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because agents use in the study may cause fetal harm.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with docetaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Response and Progression using RECIST Criteria | baseline and after two cycles of chemotherapy
  Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques (CT, MRI, x-ray) or as >10 mm with spiral CT scan.

SECONDARY OUTCOMES:
Detection of methylated and unmethylated DNA | before and after pre-operative chemotherapy (6-8 weeks)
  Treated DNA will be used for PCR using the appropriate primers. Primer sets for RUNX3 will be used for detecting methylated and unmethylated DNA. Results of methylation studies will be analysed and correlated with clinical parameters including age distribution, gender, age, staging, and treatment response. Additional genotyping may be performed on relevant polymorphisms such as XRCC, TS and CYP3A4 to correlate with treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Cassidy J, Twelves C, Van Cutsem E, Hoff P, Bajetta E, Boyer M, Bugat R, Burger U, Garin A, Graeven U, McKendric J, Maroun J, Marshall J, Osterwalder B, Perez-Manga G, Rosso R, Rougier P, Schilsky RL; Capecitabine Colorectal Cancer Study Group. First-line oral capecitabine therapy in metastatic colorectal cancer: a favorable safety profile compared with intravenous 5-fluorouracil/leucovorin. Ann Oncol. 2002 Apr;13(4):566-75. doi: 10.1093/annonc/mdf089. PMID 12056707